CLINICAL TRIAL: NCT00255918
Title: Phase 1 Trial of 3-2,4 Dimethoxbenzylidene Anabaseine in Schizophrenia
Brief Title: Investigation of the Drug Dimethoxbenzylidene Anabaseine in Treating Schizophrenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0857; R01MH061412 (NIH); DNBBS MC-R
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Evoked Potentials; 3-(2,4-dimethoxybenzylidene)anabaseine; DMXB-A; Receptors, Nicotinic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dimethoxybenzylidene anabaseine 75 mg (Experimental): Participants will take active experimental medication (Dimethoxybenzylidene anabaseine (DMXB-A) 75 mg)
  Interventions: Drug: Dimethoxybenzylidene anabaseine (DMXB-A); Drug: Placebo
- Placebo (Placebo Comparator): Participants will take placebo.
  Interventions: Drug: Dimethoxybenzylidene anabaseine (DMXB-A); Drug: Placebo
- Dimethoxybenzylidene anabaseine 150 mg (Experimental): Participants will take active experimental medication (Dimethoxybenzylidene anabaseine (DMXB-A) 150 mg)
  Interventions: Drug: Dimethoxybenzylidene anabaseine (DMXB-A); Drug: Placebo

INTERVENTIONS:
Drug: Dimethoxybenzylidene anabaseine (DMXB-A) — DMXB-A 150 mg immediate release followed by DMXB-A 75 mg 2 hours after the intiial dose
Drug: Placebo — Placebo dosed to match active medication
Drug: Dimethoxybenzylidene anabaseine (DMXB-A) — DMXB-A 75 mg immediate release followed by DMXB-A 37.5 mg 2 hours after the intiial dose

SUMMARY:
This study will determine the effectiveness of a drug, dimethoxbenzylidene anabaseine, in producing beneficial effects similar to that of nicotine in individuals with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and severe brain disorder that can significantly impact quality of life. It is characterized by delusions, paranoia, and disordered thinking. The cause of schizophrenia has not yet been determined. However, there are many treatments, including drug therapy and cognitive behavioral therapy, that may help to alleviate symptoms of the condition. Nicotinic receptors are involved in a number of biological processes; they are numerous throughout the central and peripheral nervous systems and are diverse in structure and expression. Genetic and neurobiological research has identified decreased expression of the a7 nicotinic receptor as an element in schizophrenia that is related to poor psychosocial outcome. Data indicate that drug therapy may reduce this deficit in receptor expression. Nicotine has been found to stimulate the a7 nicotinic receptor; however, the physiological dependence associated with nicotine makes it an undesirable option. Dimethoxbenzylidene anabaseine (DMXB-A) can stimulate the a7 nicotinic receptor; its advantages include easy oral administration and the lack of dependence-causing effects. This study will determine whether DMXB-A can safely and effectively stimulate the a7 nicotinic receptor in schizophrenia patients and reduce their neurobiological symptoms.

This study will last 6 weeks. Participants will have study visits each week for the duration of the study. During each visit, participants will be randomly assigned to receive either DMXB-A or placebo. An electrocardiogram (EKG) will measure the heart function of participants and participants' blood pressure will be measured. After the first dose of either DMXB-A or placebo, participants will receive a second dose 2 hours later. An evoked potential test, which measures the brain's response to stimuli, will be performed after both doses. Neuropsychological tests, such as verbal reasoning and visual retention, will be performed following the second dose of either DMXB-A or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia

Exclusion Criteria:

* History of cardiovascular illness or neurological illness other than schizophrenia
* Current substance abuse, including nicotine
* History of clozapine use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Total Scale Score for the Repeatable Battery for the Assessment of Neuropsychological Status | Measured at 2 hours after drug or placebo
  ten subtests which give five scores, one for each of the five domains tested (immediate memory, visuospatial/constructional, language, attention, delayed memory).

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale | Measured 4 hours after drug or placebo administration
  Brief Psychiatric Rating Scale (BPRS) is a rating scale used to measure psychiatric symptoms
P50 auditory evoked potential test amplitude/conditioning amplitude ratio | Measured 2.5 hours after drug or placebo administration
  The evoked response amplitude measured in mV to the initial auditory stimulus which is compared to the evoked response amplitude which is measured in mV to a second auditory stimulus that occurs 500 ms later.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado General Clinical Research Center, Denver, Colorado, United States

REFERENCES:
- [Background] Martin LF, Kem WR, Freedman R. Alpha-7 nicotinic receptor agonists: potential new candidates for the treatment of schizophrenia. Psychopharmacology (Berl). 2004 Jun;174(1):54-64. doi: 10.1007/s00213-003-1750-1. Epub 2004 Feb 19. PMID 15205879